CLINICAL TRIAL: NCT04645446
Title: A Multicenter, Randomized, Double-Masked, Placebo-Controlled Phase II Study to Evaluate the Safety and Efficacy of Pro-ocular™ 0.5% and 1% in Patients With Dry Eye Syndrome
Brief Title: Safety and Efficacy of Two Different Concentrations (0.5% and 1%) of Progesterone Topical Gel Compared to Placebo in Patients Diagnosed With Moderate to Severe Dry Eye Syndrome
Acronym: ProGIFT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 049/SI; 2019-000747-27 (EudraCT Number)
Record Dates: First submitted 2020-11-25; First posted 2020-11-27 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2021-03

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Allocation Ratio = 1:1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pro-ocular™ 1% Progesterone EP topical gel (Experimental): Multidose formulation despensing unit doses of 0.07 g of topical gel containing 0.7 mg of progesterone
  Interventions: Drug: Pro-ocular gel
- Pro-ocular™ 0.5% Progesterone EP topical gel (Experimental): Multidose formulation despensing unit doses of 0.07 g of topical gel containing 0.35 mg of progesterone
  Interventions: Drug: Pro-ocular gel
- Placebo topical gel (Placebo Comparator): Multidose formulation identical in appearance to Experimental Products despensing unit doses of 0.07 g of topical gel containing 0 mg of progesterone
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Pro-ocular gel — Topical gel in multidose formulation to be applied laterally to the forehead twice a day, morning and night for 3 months
  Arms: Pro-ocular™ 0.5% Progesterone EP topical gel; Pro-ocular™ 1% Progesterone EP topical gel
Drug: Placebo gel — Topical gel in multidose formulation to be applied laterally to the forehead twice a day, morning and night for 3 months
  Arms: Placebo topical gel

SUMMARY:
Multicenter, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group, Phase 2 clinical trial.

The study objective is to evaluate the safety and efficacy of two different concentrations (0.5% and 1%) of progesterone topical gel compared to placebo, when administered twice a day for 3 months (12 weeks) in patients diagnosed with moderate to severe dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male or female) ≥ 18 years of age.
2. Able and willing to provide voluntary written Informed Consent prior to any study related procedure.
3. Patients must be diagnosed with any type of dry eye at least 3 months before screening (Visit 0).
4. Have all the following in the same eye at Visit 0:

   * Fluorescein staining (Cornea) on NEI (National Eye Institute) grading scale > 3
   * Average Tear Film Break up Time ≤ 5 seconds
   * Schirmer Test (without anesthesia) ≥ 1 and < 10mm
5. Be able and willing to follow instructions, including participation in all study assessments and visits, according to the opinion of the investigator.

Exclusion Criteria:

1. Comorbidity with other severe or chronic conditions that in the judgment of the investigator will interfere with study assessment, such as such as glaucoma, active neuronal trigeminal disease, neuralgia.
2. Best corrected visual acuity (BCVA) baseline <20/200.
3. Condition or history other than ocular that, in the opinion of the investigator, may interfere significantly with the patient's participation in the study, such as dementia, psychosis, Parkinson's disease (interference).
4. Patient using a contact ocular lens within 7 days prior to administration of the first dose and not willing to cease using them during all study duration.
5. Female patients who are pregnant, nursing an infant, or planning a pregnancy or lactating at Screening Visit.
6. Females who are of childbearing potential and not taking adequate contraceptive precautions are excluded from the trial. Females of childbearing potential taking acceptable non-hormonal contraceptive precautions can be included (See Note A).
7. Males with partners who are pregnant or lactating or of childbearing potential and are unwilling to use condoms for the duration of the study.
8. A known adverse reaction and/or sensitivity to the study drug or its components.
9. Use of topical ocular cyclosporine, corticosteroids or any other topical anti-inflammatory treatments within 15 days prior to Visit 0 and during all study duration.
10. Routine use (more than twice a week) of a chlorinated swimming pool during the study period
11. Unwilling or unable to cease using during the study period the forbidden medications:

    * Any topical ocular ointments or gels
    * Topical and systemic glaucoma therapies
    * Systemic drugs with anticholinergic activity: anticonvulsants, antihistamines, antipsychotics, antidepressants, antimuscarinics, anti-Parkinson agents, cardiovascular agents (disopyramide), gastrointestinal agents, muscle relaxants, respiratory medications (pseudoephedrine, theophylline)
    * Lipidic artificial tears and artificial tears with preservative.
12. Unwilling to cease the use of sunscreen on the forehead or eye area during the study period.
13. Habitual cigarette smokers (tobacco, vapor cigarettes, marijuana), smoking more than 4 cigarettes per day.
14. Participation in another clinical study at the same time as the present and within 30 days prior to Visit 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining | Week 12 (Day 84) (with Last Observation Carried Forward (LOCF) imputation)
  Mean change from baseline (Visit 1 pre-dose) in corneal fluorescein staining assessed by NEI scale at Week 12 (Day 84) (with Last Observation Carried Forward (LOCF) imputation)
SANDE questionnaire | Week 12 (Day 84) (with Last Observation Carried Forward (LOCF) imputation)
  Mean change from baseline (Visit 1 pre-dose) in sum of frequency and intensity of dryness/irritation patient feeling assessed by SANDE questionnaire at Week 12 (Day 84) (with LOCF imputation)

SECONDARY OUTCOMES:
Corneal fluorescein staining | Week 12 (Day 84)
  Mean change from baseline (Visit 1 pre-dose) in corneal fluorescein staining assessed by NEI scale at Week 12 (Day 84).
SANDE questionnaire | Week 12 (Day 84)
  Mean change from baseline (Visit 1 pre-dose) in sum of frequency and intensity of dryness/irritation patient feeling assessed by SANDE questionnaire at Week 12 (Day 84).
Conjunctival fluorescein staining | Week 12 (Day 84) (with Last Observation Carried Forward (LOCF) imputation)
  Mean change from baseline (Visit 1 pre-dose) in conjunctival fluorescein staining assessed by NEI scale at Week 12 (Day 84) (with LOCF imputation).
Conjunctival fluorescein staining | Week 12 (Day 84)
  Mean change from baseline (Visit 1 pre-dose) in conjunctival fluorescein staining assessed by NEI scale at Week 12 (Day 84).
Corneal fluorescein staining | Week 2, 4, 8 (Day 14, 28, 56)
  Mean change from baseline (Visit 1 pre-dose) in corneal fluorescein staining assessed by NEI scale at Week 2, 4, 8 (Day 14, 28, 56) as intermediate study visits.
SANDE questionnaire | Week 2, 4, 8, 16 (Day 14, 28, 56,114)
  Mean change from baseline (Visit 1 pre-dose) in sum of frequency and intensity of dryness/irritation patient feeling assessed by SANDE questionnaire at Week 2, 4, 8, 16 (Day 14, 28, 56,114) as intermediate study visits.
Conjunctival fluorescein staining | Week 2, 4, 8 (Day 14, 28, 56)
  Mean change from baseline (Visit 1 pre-dose) in conjunctival fluorescein staining assessed by NEI scale at Week 2, 4, 8 (Day 14, 28, 56) as intermediate study visits.
Non-Invasive Keratograph Tear Film Break Up (NIKBUT) Time (NIKBUT) | Week 2, 4, 8, 12 (Day 14, 28, 56, 84)
  Mean change from baseline (Visit 1 pre-dose) in Non-Invasive Keratograph Tear Film Break Up Time (NIKBUT) at each applicable post-baseline visit [Week 2, 4, 8, 12 (Day 14, 28, 56, 84)].
Fluorescein Tear Film Break Up Time (TBUT) | Week 12 (Day 84)
  Mean change from baseline (Visit 1 pre-dose) in Fluorescein Tear Film Break Up Time (TBUT) at Week 12 (Day 84).
Tear meniscus height (TMH) | Week 2, 4, 8, 12 (Day 14, 28, 56, 84)]
  Mean change from baseline (Visit 1 pre-dose) in Tear meniscus height (TMH) at each applicable post-baseline visit [Week 2, 4, 8, 12 (Day 14, 28, 56, 84)].
Schirmer test | Week 4 (Day 28) and Week 12 (Day 84)
  Mean change from baseline (Visit 0 Screening) in Schirmer test at Week 4 (Day 28) and at Week 12 (Day 84).
Dry Eye-Related Quality-of-Life (DEQS) questionnaire | Each applicable post baseline visit
  Impact of dry eye on quality of life by using Dry Eye-Related Quality-of-Life (DEQS) questionnaire.
Visual Analogue Scale | Each applicable post baseline visit
  Absolute score of each symptom item in Visual Analogue Scale to each post baseline visit.
Visual Analogue Scale | Week 2, 4, 8, 12 (Day 14, 28, 56, 84)
  Mean change from baseline (Visit 1 pre-dose) in Visual Analogue Scale 7 symptoms items to each applicable post-baseline visit [Week 2, 4, 8, 12 (Day 14, 28, 56, 84)].
Corneal Sensitivity | Week 4, 12 (Day 28, 84)
  Mean change from baseline (Visit 1 pre-dose) in Corneal Sensitivity to each applicable postbaseline visit [Week 4, 12 (Day 28, 84)].
Slit Lamp Examination | Week 2, 4, 8, 12 (Day 14, 28, 56, 84)
  Mean change from baseline (Visit 0 Screening) in Slit Lamp Examination to each applicable post-baseline visit [Week 2, 4, 8, 12 (Day 14, 28, 56, 84)].

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Ospedale San Marco - Azienda Ospedaliera Universitaria, Catania
  - A.O.U. Careggi Firenze - SOD Oculistica, Florence
  - Azienda Ospedaliera Universitaria Policlinico G. Martino - UOC di Oftalmologia, Messina
  - Ospedale Luigi Sacco Polo Universitario - Oculistica, Milan